CLINICAL TRIAL: NCT02060110
Title: MADIT-CRT LONG-TERM INTERNATIONAL FOLLOW-UP REGISTRY - EUROPE
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Israeli Association for Cardiovascular Trials - IACT (Unknown)
Responsible Party: Principal Investigator, Prof. Ilan Goldenberg, MD, Director of the Israeli Association for Cardiovascular Trials, Sheba Medical Center
Other Study IDs: SHEBA-12-9492-IG-CTIL
Record Dates: First submitted 2014-02-09; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Heart Failure
Keywords: CRT; HEART FAILURE
MeSH Terms: conditions — Heart Failure | interventions — Electric Countershock

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MADIT-CRT CRT-D: Patients that were randomized to the the cardiac resynchronization therapy with defibrillation (CRT-D) device for the study
  Interventions: Device: Patients that were randomized to the the cardiac resynchronization therapy with defibrillation (CRT-D) device for the study
- MADIT-CRT ICD: Patients that were randomized to the the implantable cardioverter defibrillator (ICD) device for the study
  Interventions: Device: MADIT-CRT ICD ONLY ARM

INTERVENTIONS:
Device: Patients that were randomized to the the cardiac resynchronization therapy with defibrillation (CRT-D) device for the study
  Other Names: Boston Scientific market approved cardiac resynchronization therapy defibrillators
  Groups: MADIT-CRT CRT-D
Device: MADIT-CRT ICD ONLY ARM
  Other Names: Market approved Boston Scientific implantable cardioverter defibrillators
  Groups: MADIT-CRT ICD

SUMMARY:
The registry is designed to determine the long-term mortality and morbidity benefit as a result of Cardiac Resynchronization Therapy with Defibrillation (CRT-D) vs. Implantable Cardioverter Defibrillator (ICD) therapy in the MADIT-CRT study patient population. The registry will collect data on patients that previously participated at MADIT-CRT sites within Europe through five years of participation from their orginal enrollment in the MADIT-CRT IDE study.

ELIGIBILITY:
Inclusion Criteria:

Active patients who were enrolled in the MADIT-CRT IDE within Europe

Exclusion Criteria:

Patients who are unable or unwilling to comply with the protocol requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry involves only those patients that participated in the MADIT-CRT IDE study within Europe.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2010-05; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 36 month follow-up

SECONDARY OUTCOMES:
Heart failure event or death | 36 month follow-up
  The combined end point of heart-failure or death, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli Association for Cardiovascular Trials at Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Moss AJ, Hall WJ, Cannom DS, Klein H, Brown MW, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Higgins SL, Pfeffer MA, Solomon SD, Wilber D, Zareba W; MADIT-CRT Trial Investigators. Cardiac-resynchronization therapy for the prevention of heart-failure events. N Engl J Med. 2009 Oct 1;361(14):1329-38. doi: 10.1056/NEJMoa0906431. Epub 2009 Sep 1. PMID 19723701
- [Derived] Vidula H, Lee E, McNitt S, Polonsky B, Aktas M, Rosero S, Younis A, Solomon SD, Zareba W, Kutyifa V, Goldenberg I. Cardiac Resynchronization Therapy and Risk of Recurrent Hospitalizations in Patients Without Left Bundle Branch Block: The Long-Term Multicenter Automatic Defibrillator Implantation Trial With Cardiac Resynchronization Therapy. Circ Heart Fail. 2020 Jul;13(7):e006925. doi: 10.1161/CIRCHEARTFAILURE.120.006925. Epub 2020 Jul 1. PMID 32605387
- [Derived] Kutyifa V, Vermilye K, Solomon SD, McNitt S, Moss AJ, Daimee UA. Long-term outcomes of cardiac resynchronization therapy by left ventricular ejection fraction. Eur J Heart Fail. 2019 Mar;21(3):360-369. doi: 10.1002/ejhf.1357. Epub 2018 Dec 28. PMID 30592353
- [Derived] Sabbag A, Goldenberg I, Moss AJ, McNitt S, Glikson M, Biton Y, Jackson L, Polonsky B, Zareba W, Kutyifa V. Predictors and Risk of Ventricular Tachyarrhythmias or Death in Black and White Cardiac Patients: A MADIT-CRT Trial Substudy. JACC Clin Electrophysiol. 2016 Aug;2(4):448-455. doi: 10.1016/j.jacep.2016.03.003. Epub 2016 May 18. PMID 29759864
- [Derived] Biton Y, Kutyifa V, Cygankiewicz I, Goldenberg I, Klein H, McNitt S, Polonsky B, Ruwald AC, Ruwald MH, Moss AJ, Zareba W. Relation of QRS Duration to Clinical Benefit of Cardiac Resynchronization Therapy in Mild Heart Failure Patients Without Left Bundle Branch Block: The Multicenter Automatic Defibrillator Implantation Trial with Cardiac Resynchronization Therapy Substudy. Circ Heart Fail. 2016 Feb;9(2):e002667. doi: 10.1161/CIRCHEARTFAILURE.115.002667. PMID 26823498
- [Derived] Biton Y, Zareba W, Goldenberg I, Klein H, McNitt S, Polonsky B, Moss AJ, Kutyifa V; MADIT-CRT Executive Committee. Sex Differences in Long-Term Outcomes With Cardiac Resynchronization Therapy in Mild Heart Failure Patients With Left Bundle Branch Block. J Am Heart Assoc. 2015 Jun 29;4(7):e002013. doi: 10.1161/JAHA.115.002013. PMID 26124205
- [Derived] Daimee UA, Moss AJ, Biton Y, Solomon SD, Klein HU, McNitt S, Polonsky B, Zareba W, Goldenberg I, Kutyifa V. Long-Term Outcomes With Cardiac Resynchronization Therapy in Patients With Mild Heart Failure With Moderate Renal Dysfunction. Circ Heart Fail. 2015 Jul;8(4):725-32. doi: 10.1161/CIRCHEARTFAILURE.115.002082. Epub 2015 Jun 2. PMID 26038537
- [Derived] Goldenberg I, Kutyifa V, Klein HU, Cannom DS, Brown MW, Dan A, Daubert JP, Estes NA 3rd, Foster E, Greenberg H, Kautzner J, Klempfner R, Kuniss M, Merkely B, Pfeffer MA, Quesada A, Viskin S, McNitt S, Polonsky B, Ghanem A, Solomon SD, Wilber D, Zareba W, Moss AJ. Survival with cardiac-resynchronization therapy in mild heart failure. N Engl J Med. 2014 May 1;370(18):1694-701. doi: 10.1056/NEJMoa1401426. Epub 2014 Mar 30. PMID 24678999